CLINICAL TRIAL: NCT01784172
Title: The Efficacy and Safety Study of Electro-acupuncture for Simple Female Stress Urinary Incontinence- a Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety Study of Electroacupuncture for Simple Female Stress Urinary incontinence-a Multicenter Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Baoyan, Vice President of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012BAI24B01-2
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Stress Incontinence
Keywords: efficacy; safety; electroacupuncture; simple female stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- electroacupuncture group (Experimental): Bilateral BL33 are given acupuncture of 50～60mm with 30～45°angle to inward and downward. Bilateral B L35 are given acupuncture of 50～60mm to outward and upward. The electric stimulator is applied to bilateral BL33 and BL35.
  Every session lasts for 30 min per day. The participants are treated continuously for 6 weeks for 3 sessions a week, 18 sessions for each patient in all.
  Interventions: Device: electroacupuncture group
- sham electroacupuncture group (Experimental): Bilateral sham BL33 and sham BL35 are given sham electroacupuncture with no current output.
  Every session lasts for 30 min per day. The participants are treated continuously for 6 weeks for 3 sessions a week, 18 sessions for each patient in all.
  Interventions: Device: sham electroacupuncture group

INTERVENTIONS:
Device: electroacupuncture group — Procedure: electro-acupuncture;Points: Bilateral Zhongliao (BL33) Huiyang(BL35).Specially-made pad is stick on pierced acupoints. Bilateral BL33 are given acupuncture of 50～60mm with 30～45°angle to inward and downward by 75mm filiform needle. Bilateral BL35 are given acupuncture of 50～60mm to outward and upward by 75mm filiform needle. Twirl, lift and thrust for 3 times, until local sour and heavy feeling coming.The electric stimulator is applied to bilateral BL33 and BL35, with continuous wave,50 Hz and electric current 1- 5mA.Every session lasts for 30 min per day.The participants are treated continuously for 6 weeks for 3 sessions a week, 18 sessions for each patient in all. The treatment is designed based on recent literature research in 10 years, former result and expert consensus.
  Other Names: SDA-V electroacupuncture apparatus(Huatuo,made in China)
  Arms: electroacupuncture group
Device: sham electroacupuncture group — Procedure: sham electroacupuncture;Points: Bilateral sham Zhongliao (BL33) sham Huiyang(BL35).Specially-made pad is stick on pierced acupoints. Both sham BL33 and BL35 are given non-penetrating needling with blunt needle. Twirl, lift and thrust for 3 times. The sham electric stimulator is applied to bilateral sham BL33 and sham BL35. The mental wire has been cut off with a same outlook as the treatment group. The electric stimulator is looked normal but with no current output. Length of Treatment and the treatment sessions are the same as treatment group.
  Other Names: Sham SDZ-V electroacupuncture apparatus(Huatuo,China)
  Arms: sham electroacupuncture group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of electroacupuncture （EA） for simple female stress urinary incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is a common disease of female. The inconvenience caused by SUI affects the patients' quality of life and health seriously. To date, there has not specific therapy on SUI. Former research showed acupuncture may work for SUI. This multi-center randomized controlled clinical trial of acupuncture for simple female stress urinary incontinence is designed to confirm the efficacy and safety of EA. This project is conducted by Chinese researchers, supported by the Chinese Government. The research result is expected to provide high quality evidence of EA for simple female stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of Simple female stress urinary incontinence
* 40-75 years old
* Volunteered to join this research and signed the informed consent

Exclusion Criteria:

* urge urinary incontinence, mixed urinary incontinence, overflow urinary incontinence, etc
* After operation for urinary incontinence or pelvic floor operation
* Edeoptosis≥Degree 2
* Symptomatic urinary tract infection
* RUV>30ml
* Qmax<20ml/s
* Constrained movement of walking, stairs climbing, running
* Patients with continuous treatment for stress urinary incontinence or medicine for bladder function
* With serious cardiovascular, cerebral, liver, kidney, or psychiatric disease, diabetes, MSA, Injury of cauda equine, myeleterosis.
* During pregnancy or lactation period
* With cardiac pacemaker, Metal allergy or severe needle phobia

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
value difference of 1h pad test, compared with the baseline | the 6 weeks
  quantity of fluid loss will be measured by 1h pad test, comparing the value of 6 weeks with the baseline(0 week), the primary outcome is the value difference.

SECONDARY OUTCOMES:
average frequency difference of urinary incontinence in 72h | the 6 weeks, the15-18 weeks, 27-30 weeks
  1. The average frequency difference of urinary incontinence in 72h of the 6 weeks is the average frequency difference of urinary incontinence in 72h of 2nd, 4th, 6th weeks based on the '72h voiding diary'; 2. The average frequency difference of urinary incontinence in 72h of the15-18 weeks is the average frequency difference of urinary incontinence in 72h of 15-18 weeks based on the '72h voiding diary'; 3. The average frequency difference of urinary incontinence in 72h of the 27-30 weeks is the average frequency difference of urinary incontinence in 72h of 27-30 weeks based on the '72h voiding diary'.
ICIQ-SF | the 6, 18, 30 week
  International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) is a brief instrument used to assess the impact of UI in patients'lives
Patient subjective effectiveness evaluation | the 6, 18, 30 week
  3 point scoring: no help=0; Small help=1; Medium help=2; Great help=3
Weekly usage of pad | the 6 weeks, 7-18weeks, 19-30 weeks
  The value of 6 weeks is the average weekly usage of pads during 1-6 week; The value of 7-18weeks is the average weekly usage of pads during 7-18 weeks; The value of 19-30 weeks is the average weekly usage of pads during 19-30 weeks.
Usage of specialty therapy for Simple female stress urinary incontinence | the 6 weeks, 7-18weeks, 19-30 weeks
  Compare the difference of uase of specialty therapy for Simple female stress urinary incontinence between the 2 groups during the 1-6 weeks, 7-18 weeks and 19-30 weeks.
subgroup analysis: Relevency between 1h pad test, frequency of urinary incontinence in 72h and extent of urinary incontinence | the 6, 18, 30 week
  the 6th week: analyse the relevancy between 1h pad test and extent of urinary incontinence; the 18th and 30th weeks: analyse the relevancy between frequency of urinary incontinence in 72h and extent of urinary incontinence.
Incidence of adverse events | the 1-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Baoyan Liu, Master, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun B, Liu Y, Su T, Sun Y, Liu Z. Electroacupuncture for stress-related urinary incontinence in elderly women: data analysis from two randomised controlled studies. BMJ Support Palliat Care. 2022 May;12(e1):e164-e170. doi: 10.1136/bmjspcare-2019-002034. Epub 2020 Jan 9. PMID 31919102
- [Derived] Jiao R, Liu Y, Liu B, Liu Z. Risk factors related to acupuncture response in postmenopausal women with stress urinary incontinence: Secondary analysis of a randomized controlled trial. Medicine (Baltimore). 2019 Apr;98(16):e15220. doi: 10.1097/MD.0000000000015220. PMID 31008950
- [Derived] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Derived] Liu Z, Xu H, Chen Y, He L, Liu J, Yan S, Du R, Wu J, Liu B. The efficacy and safety of electroacupuncture for women with pure stress urinary incontinence: study protocol for a multicenter randomized controlled trial. Trials. 2013 Sep 30;14:315. doi: 10.1186/1745-6215-14-315. PMID 24079823